CLINICAL TRIAL: NCT05156294
Title: Effect of Soft Tissue Augmentation With an Acellular Dermal Matrix in Marginal Bone Levels Around Implants. A Randomized Clinical Trial
Brief Title: Effect of Soft Tissue Augmentation With an Acellular Dermal Matrix in Marginal Bone Levels Around Implants
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21/622-EC_P
Record Dates: First submitted 2021-11-11; First posted 2021-12-14 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Dental Implant Failure Nos

STUDY DESIGN:
Intervention Model Description: doubled-blind, parallel groups, randomized clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Clinical examiners evaluating and recording the outcome measurements will be masked to the treatment allocation and the patients will be asked not to reveal their treatment assignment to the examiners.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Test (Experimental): Mucoperiosteal flaps will be raised and the conventional drilling sequence for implants will be implemented (Camlog Conelog Screw-Line Promote Plus implants). Implants will be placed 1 mm below the bone crest. The diameter of the implant will be in the range of 3.8 and 4.3 mm. Consecutively, 4 to 6 mm height healing abutments and the allogenic membrane (NovoMatrix®, BioHorizon) folded in two on top of the implant (secured with the healing abutment), will be placed. Finally, flaps will be sutured with 6/0 polypropylene monofilament. Patients will be instructed to rinse with 15 ml of 0.12% chlorhexidine (Perio-Aid tratamiento, Dentaid SL, Barcelona, Spain) 60 seconds twice per day until suture removal, that will take place 14 days later. Anti-inflammatory drugs will also be prescribed (Ibuprofen 600 mg every 8 hours upon patient´s needs).
  Interventions: Device: NovoMatrix
- Control (Other): Mucoperiosteal flaps will be raised and the conventional drilling sequence for implants will be implemented (Camlog Conelog Screw-Line Promote Plus implants). Implants will be placed 1 mm below the bone crest. The diameter of the implant will be in the range of 3.8 and 4.3 mm. Finally, flaps will be sutured with 6/0 polypropylene monofilament. Patients will be instructed to rinse with 15 ml of 0.12% chlorhexidine (Perio-Aid tratamiento, Dentaid SL, Barcelona, Spain) 60 seconds twice per day until suture removal, that will take place 14 days later. Anti-inflammatory drugs will also be prescribed (Ibuprofen 600 mg every 8 hours upon patient´s needs).
  Interventions: Other: Control

INTERVENTIONS:
Device: NovoMatrix — Implants of Camlog Conelog Screw-Line Promote Plus will be placed. Implants will be placed 1 mm below the bone crest. The diameter of the implant will be in the range of 3.8 and 4.3 mm. Consecutively, 4 to 6 mm height healing abutments and the allogenic membrane (NovoMatrix®, BioHorizon) folded in two on top of the implant (secured with the healing abutment), will be placed. Finally, flaps will be sutured with 6/0 polypropylene monofilament. Patients will be instructed to rinse with 15 ml of 0.12% chlorhexidine (Perio-Aid tratamiento, Dentaid SL, Barcelona, Spain) 60 seconds twice per day until suture removal, that will take place 14 days later. Anti-inflammatory drugs will also be prescribed (Ibuprofen 600 mg every 8 hours upon patient´s needs).
  Arms: Test
Other: Control — Implants of Camlog Conelog Screw-Line Promote Plus will be placed. Implants will be placed 1 mm below the bone crest. The diameter of the implant will be in the range of 3.8 and 4.3 mm. Finally, flaps will be sutured with 6/0 polypropylene monofilament. Patients will be instructed to rinse with 15 ml of 0.12% chlorhexidine (Perio-Aid tratamiento, Dentaid SL, Barcelona, Spain) 60 seconds twice per day until suture removal, that will take place 14 days later. Anti-inflammatory drugs will also be prescribed (Ibuprofen 600 mg every 8 hours upon patient´s needs).
  Arms: Control

SUMMARY:
The main objective of this study is to evaluate the efficacy of an acellular dermal matrix membrane to increase the peri-implant soft tissue thickness and to reduce marginal bone loss during non-submerged implant placement, as compared with the standard protocol for implant placement. The test hypothesis is that placing an acellular dermal matrix membrane simultaneous to implant placement in the posterior mandible, will increase the soft tissue thickness and consequently reduce the marginal bone level changes.

The study is designed as a doubled-blind, parallel groups, randomized clinical trial with a 1-year follow-up

DETAILED DESCRIPTION:
The study is designed as a doubled-blind, parallel groups, randomized clinical trial with a 1-year follow-up. The randomization sequence will be created using a computer-generated list by an independent researcher. Allocation concealment will be kept by means of opaque sealed envelopes that will be open by one of the researchers during surgery, and revealed to the operator immediately after implant insertion.

All patients will receive standardized oral hygiene instructions consisting on the use of a manual or power-driven toothbrush and specific interdental brushes. Then, patients will be randomized to one of the following groups:

* Test Group :Mucoperiosteal flaps will be raised and the conventional drilling sequence for implants will be implemented (Camlog Conelog Screw-Line Promote Plus implants). Implants will be placed 1 mm below the bone crest. The diameter of the implant will be in the range of 3.8 and 4.3 mm. Consecutively, 4 to 6 mm height healing abutments and the allogenic membrane (NovoMatrix®, BioHorizon) folded in two on top of the implant (secured with the healing abutment), will be placed. Finally, flaps will be sutured with 6/0 polypropylene monofilament. Patients will be instructed to rinse with 15 ml of 0.12% chlorhexidine (Perio-Aid tratamiento, Dentaid SL, Barcelona, Spain) 60 seconds twice per day until suture removal, that will take place 14 days later. Anti-inflammatory drugs will also be prescribed (Ibuprofen 600 mg every 8 hours upon patient´s needs)
* Control Group: All the procedures will be the same as in the Test Group, with the only difference that no attempt to thicken the mucosa with the acellular dermal matrix will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* Periodontally healthy or with stable treated periodontitis and good oral hygiene (Full Mouth Plaque Score (FMPS) and Full Mouth Bleeding Score (FMBS) ≤ 15%, measured at six sites per tooth)
* Need for one or two implants in the posterior mandible (maximum of three missing teeth).
* Enough bone availability to place an implant with a minimum diameter of 3.8 mm and at least 7 mm length.
* Non-smoker or smokers < 10 cig/day (self-reported).
* Ability to understand the study procedures and to comply with them to the entire length of the study.

Exclusion Criteria:

* Subjects with uncontrolled systemic diseases (ASA type III).
* Subjects taking medications with immunosuppressors, bisphosphonates or high doses of corticosteroids; current drug or alcohol use or dependence that could interfere with adherence to study requirements.
* Pregnant or lactating women.
* Allergy to collagen or analgesics/anti-inflammatory non-steroid drugs.
* History of cancer requiring radiotherapy or chemotherapy during the last 5 years.
* Local inflammation (including untreated periodontitis)
* Severe bruxism or clenching habits.
* Any kind of bone augmentation performed on the implant site, with a healing period <6 months
* Less than 4 mm of keratinized mucosa
* Post-extraction sites with <12 weeks of healing
* Lack of primary implant stability assessed intrasurgically.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Change in marginal alveolar crest | 1 year
  The primary outcome variable of this trial is the change in the marginal alveolar crest after the surgical intervention, assessed by the radiographic change of interproximal bone levels. It will be assessed with periapical radiographs, immediately after surgery and at 6 months and 12 months after loading, by means of computer image analysis software (Image J, National Institute of Health [NIH], Bethesda, Maryland). The calibration of the periapical radiographs will be performed using the distance between two implant threads or the length of the implant.

SECONDARY OUTCOMES:
Duration of surgical intervention. | from the tooth extraction to the end of the surgery
  Will be measured using the stopwatch, starting from the tooth extraction and ending with the suturing
Wound healing | After a week
  Will be assessed using Landry index
Change of keratinized tissue width | 1 year
  Will be measured from the soft tissue margin to the muco-gingival junction at the mid-buccal aspect.
Change in peri-implant soft tissue thickness | 1 year
  Expressed in millimeters, measured by linear and volumetric analysis. The STL's representing the tissue contours at baseline, 2 months (M), 6M and 12M, will be superimposed to the DICOM files representing the hard tissue at baseline and 12M.
Change of the peri-implant soft tissue health | 1 year
  Will be measured in six points at the implant of interest, using a University of North Carolina (UNC-15) periodontal probe.
Interproximal recession | 1 year
  Will be measured as the distance in mm between the peak of the papilla and the incisal edge.
Full-mouth plaque and bleeding scores | 1 year
  as the percentage of total surfaces (four aspects per tooth) that revealed plaque (Full mouth plaque score or FMPS, O'Leary et al., 1972) and bleeding on probing, respectively.
  Absence or presence of plaque on each surface in the dentition will be recorded in dichotomous manner, with subsequent calculation of the full-mouth plaque score as percentage of the surfaces with plaque to the total number of surfaces assessed; similarly, full-mouth bleeding score will be calculated, assessing presence of bleeding upon gentle probing with standardized force of 0.25 Newtons (N).
Patient-reported outcome measures for pain and discomfort | 14 days
  will be reported by assessing post-surgical morbidity and patient-reported experience measures (Tonetti et al., 2018); Patients will be instructed to use a post-operative diary for the first 14 days after the surgery to capture patient-reported experience measures.
  The diary will be designed to assess patient recovery in four main areas: post-surgery sequelae, pain and discomfort, oral function and interference with daily activities. Patient perception of pain and discomfort will be rated using a Visual Analogue Scale (VAS) scale. Patients will be asked to report the number of tablets and days taken as painkillers or anti-inflammatory drugs.
Patient Global Assessment | 1 year
  Apart from that, patient perception of the difficulty of surgical intervention, patient perception of pain during the procedure and patient preference for alternate therapy will be recorded at the end of the surgery, using the VAS scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Mad, Spain

REFERENCES:
- [Background] Canullo L, Fedele GR, Iannello G, Jepsen S. Platform switching and marginal bone-level alterations: the results of a randomized-controlled trial. Clin Oral Implants Res. 2010 Jan;21(1):115-21. doi: 10.1111/j.1600-0501.2009.01867.x. PMID 20070752
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Background] Linkevicius T, Puisys A, Steigmann M, Vindasiute E, Linkeviciene L. Influence of Vertical Soft Tissue Thickness on Crestal Bone Changes Around Implants with Platform Switching: A Comparative Clinical Study. Clin Implant Dent Relat Res. 2015 Dec;17(6):1228-36. doi: 10.1111/cid.12222. Epub 2014 Mar 28. PMID 24673875